CLINICAL TRIAL: NCT02864316
Title: Phase 2 Study of Nivolumab in Solid Tumors Induced by Prior Radiation Exposure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1695; IRB00105682 (Other: JHMIRB)
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumors Induced by Prior Radiation Exposure
Keywords: radiation-induced solid tumors; Nivolumab; Phase 2 study
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation-Induced Metastatic Sarcoma (Experimental): a flat dose of Nivolumab 240 mg will be administered intravenously every 2 weeks until disease progression.
  Interventions: Drug: Nivolumab
- Radiation-Induced Non-Sarcoma Metastatic Solid Tumors (Experimental): a flat dose of Nivolumab 240 mg will be administered intravenously every 2 weeks until disease progression.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558; MDX-1106

SUMMARY:
The purpose of this study is to determine whether Nivolumab is effective in the treatment of radiation-induced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable solid tumor which standard curative or palliative measures do not exist or are no longer effective. The primary site of the metastatic or unresectable tumor must have arisen within a previously irradiated site and be considered a radiation-induced tumor.
* Pre-treatment tumor specimen available. Patients with no available archived specimen must be willing to undergo a pre-treatment tumor biopsy.
* Measurable disease.
* Progressive disease on study entry.
* Received adjuvant or neoadjuvant chemotherapy and developed recurrent or metastatic disease within 6 months of completing therapy.
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Life expectancy of greater than 3 months.
* Adequate organ and marrow function as defined below:
* White Blood Cell >2,000/per microliter
* Absolute neutrophil count >1,500/per microliter
* Platelets >100,000/per microliter
* Hemoglobin ≥9.0 g/dL
* Total bilirubin ≤1.5 times the institutional upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate Aminotransferase(SGOT)/Alanine Aminotransferase (SGPT) <3 X institutional ULN
* Creatinine ≤1.5 X institutional ULN OR
* Creatinine clearance >40 mL/min for patients with creatinine Levels above institutional normal (calculated using the Cockcroft-Gault formula below)
* Female Creatinine Clearance = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
* Male Creatinine Clearance = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
* Women of childbearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry and for the duration of study participation and up to 31 weeks after the last dose of nivolumab.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of nivolumab.
* Ability to understand and the willingness to sign a written informed consent document.
* Biopsiable disease at the time of enrollment as biopsies after progression are required for participation.

Exclusion Criteria:

* Any active, known or suspected autoimmune disease.
* Requiring continuous supplemental oxygen.
* Chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or unresolved toxicity due to agents administered more than 2 weeks earlier.
* Uncontrolled brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab.
* Uncontrolled inter-current illness.
* Pregnant or currently breastfeeding.
* Receiving any other anticancer therapy.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA- 4 antibody therapies, any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
* History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating ongoing acute or chronic infection.
* Requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Forde, MB, BCH, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Cancer Center @ Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects were screen failures
Groups:
- Radiation-Induced Metastatic Sarcoma; Radiation-Induced Non-Sarcoma Metastatic Solid Tumors: a flat dose of Nivolumab 240 mg will be administered intravenously every 2 weeks until disease progression.
  Nivolumab
Period: Overall Study
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Progressive Disease | 2 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate
Description: Number of participants with response. Response will be assessed at baseline (within 4 weeks prior to starting nivolumab) and then every 8 weeks while on Nivolumab, up to 24 weeks. The best objective response will be assessed at 24 weeks. Response will be defined based on RECIST 1.1 criteria where complete response (CR)= disappearance of all target lesions, partial response (PR) is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: Up to 24 weeks
Population: Data was not collected for 1/2 participants from the non-sarcoma arm since the participant was discontinued from therapy (due to adverse event) before disease re-evaluation for response could be performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 2 | 1
Participants
  PD | 2 | 1
  SD | 0 | 0
  PR | 0 | 0
  CR | 0 | 0

2. Secondary Outcome: Percentage of Patients Progression-free at 24 Weeks From the Time of Enrollment
Description: Disease status at 24 weeks will be compared to disease status at the time of enrollment, and response coded based on RECIST 1.1 criteria.
Time Frame: 24 weeks
Population: Data was not collected to assess this outcome measure since no participants remained on the study at 24 weeks.
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Number of participants alive without progression.
Time Frame: Up to 22 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, accessed up to 3 years.
Time Frame: Up to 22 months
Population: Data was not collected to assess this outcome measure since none of the participants experienced a response.
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants with treatment-related adverse events as defined by CTCAE 4.0 criteria.
Time Frame: up to 100 days post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

6. Secondary Outcome: Overall Survival
Description: Overall survival was planned to be measured at 5 years post-intervention as the time from enrollment until death. Instead, due to early termination for low accrual, the number of participants alive at the time of study termination is reported.
Time Frame: Up to 22 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 100 days after last-dose of therapy
Arm/Group | Radiation-Induced Metastatic Sarcoma | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation-Induced Metastatic Sarcoma (N=2) | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors (N=2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation-Induced Metastatic Sarcoma (N=2) | Radiation-Induced Non-Sarcoma Metastatic Solid Tumors (N=2)
Hyperhhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Edema - limbs (General disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT02864316/Prot_SAP_000.pdf